CLINICAL TRIAL: NCT00797745
Title: A Study of SCH 900518 in Previously Untreated Subjects With Genotype 1 Chronic Hepatitis C (Protocol No. P05104)
Brief Title: A Pharmacokinetics/Pharmacodynamics Study of SCH 900518 in Previously Untreated Subjects With Genotype 1 Chronic Hepatitis C (Protocol No. P05104AM2)(COMPLETED)
Acronym: NEXT-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05104
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Hepatitis C, Chronic
Keywords: genotype 1 infection
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin; narlaprevir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Standard of Care (Active Comparator): PegIntron 1.5 mcg/kg SC weekly plus ribavirin 600 to 1400 mg daily (weight-based) by mouth twice daily for 48 weeks.
  * Subjects with >= 1 log decrease from baseline in HCV-RNA levels after 12 weeks, but still above the lower limit of quantitation, have the option of crossing over to PegIntron, ribavirin plus SCH 900518 400 mg and ritonavir 100 mg daily for 12 weeks. This is followed by standard of care, PegIntron and ribavirin, for a total treatment duration of up to 48 weeks.
  Interventions: Biological: peginterferon alfa 2b; Drug: ribavirin; Drug: SCH 900518; Drug: ritonavir
- 2 (Experimental): PegIntron 1.5 mcg/kg SC weekly plus ribavirin 600 to 1400 mg daily (weight-based) by mouth twice daily plus SCH 900518 200 mg daily plus ritonavir 100 mg daily for 12 weeks. Depending on HCV-RNA levels after 4 weeks of SCH 900518, patients will receive an additional 12 or 36 weeks of PegIntron/ribavirin. Total treatment duration will be 24 or 48 weeks.
  Interventions: Biological: peginterferon alfa 2b; Drug: ribavirin; Drug: SCH 900518; Drug: ritonavir
- 3 (Experimental): PegIntron 1.5 mcg/kg SC weekly plus ribavirin 600 to 1400 mg daily (weight-based) by mouth twice daily plus SCH 900518 400 mg daily plus ritonavir 100 mg daily for 12 weeks. Depending on HCV-RNA levels after 4 weeks of SCH 900518, patients will receive an additional 12 or 36 weeks of PegIntron/ribavirin. Total treatment duration will be 24 or 48 weeks.
  Interventions: Biological: peginterferon alfa 2b; Drug: ribavirin; Drug: SCH 900518; Drug: ritonavir
- 4 (Experimental): 4 week lead-in with PegIntron 1.5 mcg/kg SC weekly plus ribavirin 600 to 1400 mg daily (weight-based) by mouth twice daily followed by PegIntron plus ribavirin plus SCH 900518 200 mg daily plus ritonavir 100 mg daily for 12 weeks. Depending on HCV-RNA levels after 4 weeks of SCH 900518, patients will receive an additional 8 or 32 weeks of PegIntron/ribavirin. Total treatment duration will be 24 or 48 weeks.
  Interventions: Biological: peginterferon alfa 2b; Drug: ribavirin; Drug: SCH 900518; Drug: ritonavir
- 5 (Experimental): 4 week lead-in with PegIntron 1.5 mcg/kg SC weekly plus ribavirin 600 to 1400 mg daily (weight-based) by mouth twice daily followed by PegIntron plus ribavirin plus SCH 900518 400 mg daily plus ritonavir 100 mg daily for 12 weeks. Depending on HCV-RNA levels after 4 weeks of SCH 900518, patients will receive an additional 8 or 32 weeks of PegIntron/ribavirin. Total treatment duration will be 24 or 48 weeks.
  Interventions: Biological: peginterferon alfa 2b; Drug: ribavirin; Drug: SCH 900518; Drug: ritonavir
- 6 (Experimental): PegIntron 1.5 mcg/kg SC weekly plus ribavirin 600 to 1400 mg daily (weight-based) by mouth twice daily plus SCH 900518 100 mg twice daily plus ritonavir 100 mg twice daily for 12 weeks. Depending on HCV-RNA levels after 4 weeks of SCH 900518, patients will receive an additional 12 or 36 weeks of PegIntron/ribavirin. Total treatment duration will be 24 or 48 weeks.
  Interventions: Biological: peginterferon alfa 2b; Drug: ribavirin; Drug: SCH 900518; Drug: ritonavir
- 7 (Experimental): 4 week lead-in with PegIntron 1.5 mcg/kg SC weekly plus ribavirin 600 to 1400 mg daily (weight-based) by mouth twice daily followed by PegIntron plus ribavirin plus SCH 900518 600 mg daily plus ritonavir 100 mg daily for 12 weeks. Depending on HCV-RNA levels after 4 weeks of SCH 900518, patients will receive an additional 8 or 32 weeks of PegIntron/ribavirin. Total treatment duration will be 24 or 48 weeks.
  Interventions: Biological: peginterferon alfa 2b; Drug: ribavirin; Drug: SCH 900518; Drug: ritonavir

INTERVENTIONS:
Biological: peginterferon alfa 2b — 1.5 mcg/kg subcutaneously weekly for up to 24 or 48 weeks
  Other Names: PegIntron
Drug: ribavirin — ribavirin 600 to 1400 mg daily (weight-based dosing) by mouth twice daily for up to 24 or 48 weeks
  Other Names: REBETOL
Drug: SCH 900518 — SCH 900518 100 mg tablets taken as 200 mg PO QD, 100 mg PO BID, 400 mg PO QD, or 600 mg PO QD for 12 weeks.
Drug: ritonavir — Ritonavir 100 mg capsules taken as 100 mg PO QD or 100 mg PO BID for 12 weeks.
  Other Names: Norvir

SUMMARY:
SCH 900518 is a potent oral inhibitor of HCV NS3 protease which disrupts hepatitis C virus (HCV) polyprotein processing. SCH 900518, when added to the current standard of care (SOC), peginterferon-alfa plus ribavirin, would likely increase the proportion of patients achieving undetectable HCV-RNA levels and sustained virologic response (SVR). In this study, SCH 900518 would be used in combination with low doses of ritonavir to enhance the levels of SCH 900518 within the body and reduce the number of daily SCH 900518 tablets required. The purpose of this study is to identify the optimal dose and schedule (once or twice a day) of SCH 900518 plus ritonavir in previously untreated patients with genotype 1 chronic hepatitis C when given in combination with SOC. The study compares SOC to 6 experimental arms. In the experimental arms, SOC plus SCH 900518 doses of 200, 400 and 600 mg once daily or 100 mg twice daily with ritonavir 100 mg once or twice daily will be explored. The benefits of a 4 week lead-in with PegIntron and ribavirin prior to the addition of SCH 900518 will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with CHC HCV genotype 1 with no previous treatment for CHC
* 18 to 55 years of age
* Weight between 40 and 125 kg
* Previously documented CHC genotype 1 infection
* Liver biopsy within 2 years of Screening with histology consistent with chronic hepatitis C and no evidence of bridging fibrosis or cirrhosis
* Subject and subject's partner(s) must each agree to use acceptable methods of contraception for at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study drug
* Subjects must be willing to give written informed consent

Exclusion Criteria:

* Prior treatment for hepatitis C other than herbal remedies
* HIV positive or known to be co-infected with hepatitis B
* Medically significant gallbladder or hepatobiliary findings on Screening ultrasound
* Use of any known significant inducers or substrates of CYP3A4 two weeks prior to start of study medications
* Use of herbal supplements (Milk Thistle permitted)
* Diabetic and hypertensive subjects with clinically significant ocular examination findings
* Current moderate or severe depression
* History of depression associated with any of the following:

  * Hospitalization for depression
  * Electroconvulsive therapy for depression.
  * Depression that resulted in a prolonged absence from work and/or significant disruption of daily functions
* Suicidal or homicidal ideation and/or attempt
* History of severe psychiatric disorders
* Past history or current use of lithium
* Clinical diagnosis of substance abuse of alcohol, intravenous drugs, inhalational (not including marijuana), psychotropics, narcotics, cocaine use, prescription or over-the-counter drugs within 5 years of Day 1
* Past or current use of opiate agonist substitution therapy
* Any known pre-existing medical condition (CNS, cardiac, pulmonary, immune mediated) that could interfere with the subject's participation in and completion of the study
* Active clinical gout within the last year
* Hemoglobinopathy or coagulopathy
* Myelodysplastic syndromes
* Organ transplants other than cornea and hair
* Poor venous access that precludes routine peripheral blood sampling or an indwelling venous catheter
* Subjects with a history of gastric surgery (eg, stapling, banding, bypass) or subjects with a history of malabsorption disorders (eg, celiac sprue disease)
* Evidence of active or suspected malignancy, or a history of malignancy, within the last 5 years (except adequately treated basal cell carcinoma of the skin). Subjects under evaluation for malignancy are not eligible.
* Subjects who are pregnant or nursing
* Subjects who intend to become pregnant during the study period
* Male subjects with partners who are, or intend to become, pregnant during the study period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the proportion of subjects with undetectable HCV-RNA after 4 weeks of treatment with SCH 900518. | After 4 weeks of treatment with SCH 900518

SECONDARY OUTCOMES:
Rate of viral decline during the first 4 weeks of dosing with SCH 900518 | After 4 and 12 weeks of treatment with SCH 900518, at EOT and FW 24
Proportion of subjects with undetectable HCV-RNA at both 4 and 12 weeks of dosing with SCH 900518 | After 4 and 12 weeks of treatment with SCH 900518, at EOT and FW 24
Proportion of subjects with undetectable HCV-RNA at end of treatment (EOT) and follow-up week 24 (FW24) | After 4 and 12 weeks of treatment with SCH 900518, at EOT and FW 24